CLINICAL TRIAL: NCT05077631
Title: A Phase I, Double-Blind, Placebo-controlled, Randomized Study to Evaluate the Effects of Single Ascending Oral Doses of ACD856 on Safety, Tolerability and Pharmacokinetics in Healthy Adults
Brief Title: Study to Evaluate the Effects of Single Ascending Oral Doses of ACD856 on Safety, Tolerability and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlzeCure Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2000CI-001
Record Dates: First submitted 2021-04-01; First posted 2021-10-14 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease; Cognition Disorder
Keywords: Cognition Disorder; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACD856 (Experimental)
  Interventions: Drug: ACD856; Drug: ACD856 (fed cohort)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACD856 — Single oral doses of ACD856 administered in a fasted state in escalation schedule of dose 1, dose 2, dose 3, dose 4, dose 5, dose 6 and dose 7. The escalation schedule may be adapted based on evaluation by internal Safety Review Committee.
  Arms: ACD856
Drug: Placebo — Placebo oral solution
  Arms: Placebo
Drug: ACD856 (fed cohort) — Single oral dose of ACD856 in fed state of either dose 4 or dose 5.
  Arms: ACD856

SUMMARY:
The SAD design of the study is based on the aim to study safety, tolerability and PK of selected doses of ACD856 in a limited number of healthy volunteers. ACD856 will be administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to any study-mandated procedure.´
* Willing and able to comply with study requirements.
* Healthy males and healthy women of non-childbearing potential aged ≥18 and <65 years at screening.
* BMI ≥18.0 and ≤30.0 kg/m2 at screening.
* Males and females of non-childbearing potential may be included in the study. Male subjects must be willing to use condom or be vasectomized or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of dosing until 3 months after dosing with the IMP.
* Clinically acceptable medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.

Exclusion Criteria:

* Planned treatment or treatment with another investigational drug within 3 months prior to randomization.
* Positive screen for drugs of abuse or a positive alcohol result at screening or admission to the clinic.
* Clinically relevant findings in laboratory parameters, ECG or vital signs at screening
* Current smokers or users of nicotine products.
* History of alcohol abuse or excessive intake of alcohol.
* Presence or history of drug abuse.
* History of, or current use of, anabolic steroids.
* Excessive caffeine consumption.
* Plasma donation within one month of screening or blood donation prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) | 8 days
  Number of subjects and percentage of subjects with AEs
Clinically significant changes in 12-lead ECGs | 8 days
  Number of subjects and percentage of subjects with clinically significant changes in 12-lead ECGs
Clinically significant changes in vital signs | 8 days
  Number of subjects and percentage of subjects with clinically significant changes in vital signs or stool frequency
Clinically significant changes in hematology, clinical chemistry, coagulation and/or urinalysis parameters | 8 days
  Number of subjects and percentage of subjects with clinically significant changes in any safety laboratory assessments.
Clinically significant changes in physical examinations | 8 days
  Number of subjects and percentage of subjects with clinically significant changes in physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sandin, Study Director — AlzeCure Pharma
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson B, Bylund J, Halldin MM, Rother M, Rein-Hedin E, Onnestam K, Segerdahl M. ACD856, a novel positive allosteric modulator of Trk receptors, single ascending doses in healthy subjects: Safety and pharmacokinetics. Eur J Clin Pharmacol. 2024 May;80(5):717-727. doi: 10.1007/s00228-024-03645-1. Epub 2024 Feb 14. PMID 38353689